CLINICAL TRIAL: NCT04184297
Title: Effectiveness and Safety of Maintenance Treatment With Combination of Tiotropium and Olodaterol in Comparison to Maintenance Treatment With a Combination of Inhaled Corticosteroids, Long-acting β2 Agonists and Long-acting Muscarinic Antagonists in COPD Patients
Brief Title: Comparative Effectiveness and Safety of Tiotropium and Olodaterol in Comparison to Triple Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0094
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects initiated with Tiotropium and Olodaterol (Tio+Olo)
  Interventions: Drug: Tiotropium and Olodaterol (Tio+Olo)
- Subjets initiated with LABA/LAMA/ICS: Long-acting beta2/ Long-acting muscarinic antagonists/Inhaled corticosteriods
  Interventions: Drug: Long-acting beta2-agonist and Inhaled corticosteroids (LABA and ICS)

INTERVENTIONS:
Drug: Tiotropium and Olodaterol (Tio+Olo) — drug
  Groups: Subjects initiated with Tiotropium and Olodaterol (Tio+Olo)
Drug: Long-acting beta2-agonist and Inhaled corticosteroids (LABA and ICS) — drug
  Groups: Subjets initiated with LABA/LAMA/ICS

SUMMARY:
To assess the comparative effectiveness of combination Tiotropium and Olodaterol (Tio+Olo) (FDC) compared to combination LAMA/LABA and ICS (fixed or open), and to explore whether this varies across COPD sub populations defined by exacerbation risk

ELIGIBILITY:
Inclusion Criteria:

* New users of Tio+Olo on the same date or of LABA, LAMA and ICS, either as a fixed-dose combination (LABA/LAMA/ICS) or free combination (LABA/ICS + LAMA, etc), on the same date between January 2013 and March 2019.
* Diagnosis of COPD prior to first maintenance inhaler and age ≥ 40 years at index date

Exclusion Criteria:

* Less than one year of medical history information prior to the date of combined treatment initiation (index date)
* Lung cancer, interstitial lung disease, or lung transplantation at any time prior to the index date
* Asthma diagnosis within one year prior to the index date

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD inititated with Tio+Olo in comparison to patients treated with ICS/LABA/LAMA
Sampling Method: Non-Probability Sample
Enrollment: 27190 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HealthCore, Inc., Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study investigate the effectiveness and safety of maintenance treatment with combination of tiotropium and olodaterol comparing to maintenance treatment with combination of inhaled corticosteroids in patients with chronic obstructive pulmonary disease (COPD) based on existing data.
Pre-assignment Details: The study was conducted using existing administrative healthcare claims and laboratory result data captured in the HealthCore Integrated Research Database (HIRD). The observation period was from January 2013 until the most recent date available at the time that the cohort is extracted (March 2019).
Groups:
- Tiotropium+Olodaterol: All patients in the HealthCore Integrated Research Database (HIRD) with a diagnosis of Chronic obstructive pulmonary disease (COPD) who received combination Tiotropium+Olodaterol (Tio + Olo) treatment from 1 January 2013 until 31 March 2019.
- LABA/LAMA/ICS: All patients in the HealthCore Integrated Research Database (HIRD) with a diagnosis of Chronic obstructive pulmonary disease (COPD) who received combination Long-acting beta2-agonist (LABA) / Long-acting muscarinic antagonists (LAMA) / Inhaled corticosteroids (ICS) treatment from 1 January 2013 until 31 March 2019.
Period: Overall Study
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS
Started | 2864 | 24326
Completed | 2864 | 24326
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) from HealthCore Integrated Research Database (January 2013 - March 2019) that meet all inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS | Total
Number analyzed (Participants) | 2864 | 24326 | 27190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (10.5) | 66.8 (10.7) | 66.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1349 | 11701 | 13050
  Male | 1515 | 12625 | 14140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Incidence rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbation was reported. Time to the first Chronic obstructive pulmonary disease (COPD) exacerbation will be measured from cohort entry until the occurrence of a hospitalization for COPD (severe exacerbation) or Emergency Department (ED) visit for COPD with the prescription of an antibiotic and/or an oral corticosteroid on the same day (moderate exacerbation).
Time Frame: From cohort entry (index date) until the occurrence of a hospitalization for COPD (severe exacerbation), ED visit for COPD or prescription of an antibiotic and oral corticosteroid on the same day (moderate exacerbation). Up to 1 year after cohort entry.
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) from HealthCore Integrated Research Database (January 2013 - March 2019) that meet all inclusion criteria, with laboratory result data available and non-missing endpoint outcomes.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS
Number analyzed (Participants) | 2864 | 24326
Events per 1000 person-days | 1.32 [1.19 to 1.48] | 1.14 [1.10 to 1.18]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol vs LABA/LAMA/ICS; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid (LABA/LAMA/ICS) therapy combination on the risk of first COPD exacerbation for overall population; Test type: Other; Regression, Cox; The method was used to calculate hazard ratios with 95% confidence intervals; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.76 to 0.96] — Hazard ratio of Tiotropium+Olodaterol versus LABA/LAMA/ICS

2. Secondary Outcome: Overall Incidence Rate of Hospitalization for Community-acquired Pneumonia (Serious Pneumonia)
Description: Overall incidence rate of first hospitalization for community-acquired pneumonia (serious pneumonia).
Time Frame: From cohort entry (index date) until the occurrence of hospitalization for community-acquired pneumonia (serious pneumonia). Up to 1 year after cohort entry.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS
Number analyzed (Participants) | 2864 | 24326
Events per 1000 person-days | 0.25 [0.20 to 0.32] | 0.24 [0.22 to 0.25]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol vs LABA/LAMA/ICS; Cox proportional hazard regression models were used to assess the effect of Tiotropium + Olodaterol combination versus the Long-acting beta agonist / inhaled corticosteroid (LABA/LAMA/ICS) therapy combination on the risk of a hospitalization for community-acquired pneumonia for overall population; Test type: Other; Regression, Cox; This method was used to calculate hazard ratios with 95% confidence intervals; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.64 to 1.07] — Hazard ratio of Tiotropium+Olodaterol versus LABA/LAMA/ICS

3. Primary Outcome: Incidence Rate of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation - Without Exacerbation Within 30 Days Prior to Cohort Entry
Description: Incidence rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbation excluding participants who had exacerbation within 30 days prior to cohort entry, was reported. Time to the first Chronic obstructive pulmonary disease (COPD) exacerbation will be measured from cohort entry until the occurrenceof a hospitalization for COPD (severe exacerbation) or Emergency Department (ED) visit for COPD with the prescription of an antibiotic and/or an oral corticosteroid on the same day (moderate exacerbation).
Time Frame: as for outcome 1
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) from HealthCore Integrated Research Database (January 2013 - March 2019) that meet all inclusion criteria, and non-missing endpoint outcomes. Participants with exacerbation within 30 days prior to cohort entry were excluded.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-days
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS
Number analyzed (Participants) | 2591 | 18352
Events per 1000 person-days | 1.18 [1.05 to 1.33] | 0.99 [0.95 to 1.03]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol vs LABA/LAMA/ICS; [analysis description as in outcome 1, analysis 1]; Test type: Other; Regression, Cox; The method was used to calculate hazard ratios with 95% confidence intervals; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.91 to 1.19] — Hazard ratio of Tiotropium+Olodaterol versus LABA/LAMA/ICS

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data retrieved from HealthCore Integrated Research Database (HIRD) database, safety monitoring and safety reporting on an individual case level is not applicable. Total number of participants at risk is 0 since adverse events were not planned to be collected and reported for this study.
Arm/Group | Tiotropium+Olodaterol | LABA/LAMA/ICS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT04184297/Prot_SAP_000.pdf